CLINICAL TRIAL: NCT03679481
Title: The Effect of Tranexamic Acid on Blood Loss and Transfusion Requirements Following Open Femur Fracture Surgery
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: study not started due to lack of funding
Sponsor: The University of Texas Health Science Center, Houston (Other)
Responsible Party: Principal Investigator, Stephen Warner, Assistant Professor, The University of Texas Health Science Center, Houston
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: HSC-MS-17-0920
Record Dates: First submitted 2018-07-24; First posted 2018-09-20 (Actual); Last update posted 2019-10-17 (Actual); Status verified 2019-10

CONDITIONS: Blood Loss Following Open Femur Fracture Surgery
MeSH Terms: interventions — Tranexamic Acid; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Tranexamic acid (TXA) (Experimental): Following induction of anesthesia and prior to surgical incision, patients will receive 1 gram of intravenous TXA mixed in 100cc of normal saline.
  Interventions: Drug: Tranexamic acid (TXA)
- Normal saline (Placebo Comparator): Following induction of anesthesia and prior to surgical incision, patients will receive 100cc of normal saline.
  Interventions: Drug: Normal saline

INTERVENTIONS:
Drug: Tranexamic acid (TXA) — Following induction of anesthesia and prior to surgical incision, patients will receive 1 gram of intravenous TXA mixed in 100cc of normal saline.
  Arms: Tranexamic acid (TXA)
Drug: Normal saline — Following induction of anesthesia and prior to surgical incision, patients will receive 100cc of normal saline.
  Arms: Normal saline

SUMMARY:
The purpose of this study is to determine the effect of tranexamic acid (TXA) on blood loss and transfusion requirements in patients with femur fractures requiring open surgical approaches.

ELIGIBILITY:
Inclusion Criteria:

* Patients admitted to Memorial Hermann Medical Center with acute femur fractures that require open surgical approaches for fracture reduction and implant application, including patients with subtrochanteric, high-energy intertrochanteric, periprosthetic, and intra-articular distal femur fractures.

Exclusion Criteria:

* Preoperative use of any anticoagulant
* History of deep venous thrombosis or pulmonary embolus
* Allergy to TXA
* Hepatic dysfunction (AST/ALT > 60)
* Renal dysfunction (Cr > 1.5 or GFR < 30)
* History of cerebrovascular accident in the past 12 months
* Active coronary artery disease (event in the past 12 months)
* Presence of drug-eluting stent
* Color blindness
* Presence of an additional acute injury that could contribute to blood transfusion requirements

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2020-04-01 (Estimated); Primary Completion 2021-04-01 (Estimated); Study Completion 2021-04-01 (Estimated)

PRIMARY OUTCOMES:
Transfusion requirements as assessed by number of packed red blood cell units received | from the time of surgery to hospital discharge (about 3-5 days)

SECONDARY OUTCOMES:
Surgical blood loss as assessed by change in red blood cell volume | baseline, while in PACU (which is about 4-6 hours after surgery)
  Blood loss will be determined using the following calculations:
  [Patient's Blood Volume (PBV) = (k1 x Height^3 (m)) + (k2 x Weight (kg)) + k3] (- k1 = 0.3669, k2 = 0.03219, and k3 = 0.6041 for men) (- k1 = 0.3561, k2=0.03308, and k3 = 0.1833 for women)
  Multiplying the PBV by the hematocrit (Hct) gives the red blood cell (RBC) volume. As such, a change in the RBC volume can be calculated from a change in the Hct level as follows. PACU is post-anesthesia care unit: [Operative RBC volume loss = PBV x (Day of surgery Hct - PACU Hct)]
  If a patient requires an intraoperative transfusion, the calculation will be adjusted as follows:
  Operative RBC volume loss = [ [PBV x (Day of surgery Hct - PACU Hct)] +)] + (No. of Units Transfused x 0.285) / (Day of surgery Hct - Post-op Hct) / 2) ]
Surgical blood loss as assessed by an intraoperative cell salvage machine | at the time of surgery
  The intraoperative cell salvage machine allows for a precise estimation of surgical blood loss.
Length of hospital stay | from the time of hospital admission to the time of hospital discharge (about 5 days)
Number of participants with complications | 6 weeks after surgery
  Complications include infection, venous thromboembolic event, and mortality.

CONTACTS AND LOCATIONS:
Overall Officials: Stephen J Warner, MD, PhD, Principal Investigator — The University of Texas Health Science Center, Houston